CLINICAL TRIAL: NCT07112859
Title: Evaluation of Success of Complete Pulpotomy With Biodentine on Mature Permanent Single Rooted Teeth With Symptomatic Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Farhana Altaf, Dr Farhana, HITEC-Institute of Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dr Farhana altaf
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — tricalcium silicate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complete Pulpotomy with Biodentine (Experimental): Patients with mature permanent single-rooted teeth diagnosed with symptomatic irreversible pulpitis will undergo complete pulpotomy. The coronal pulp will be removed, and Biodentine will be placed on the remaining radicular pulp, followed by restoration. Patients will be followed up to evaluate treatment success.
  Interventions: Procedure: Complete Pulpotomy with Biodentine

INTERVENTIONS:
Procedure: Complete Pulpotomy with Biodentine — Administration of local anesthesia followed by rubber dam isolation.
  Removal of coronal pulp tissue to perform a complete pulpotomy.
  Hemostasis achieved with saline-soaked cotton pellet.
  Placement of Biodentine as the pulp-capping agent on the radicular pulp.
  Temporary restoration placed immediately after Biodentine placement.
  Permanent composite restoration placed after 1 week.
  Follow-up visits at 7 days, 1 month, and 3 months for clinical and radiographic evaluation.

SUMMARY:
This study aims to evaluate the clinical success of complete pulpotomy using Biodentine in mature permanent single-rooted teeth diagnosed with symptomatic irreversible pulpitis. Complete pulpotomy involves removal of the coronal pulp and preservation of radicular pulp vitality using a biocompatible pulp-capping material. Biodentine, a calcium silicate-based cement, has favorable biological properties, including biocompatibility, antibacterial effects, and dentin bridge formation potential. A total of 84 patients meeting the inclusion criteria will be enrolled and treated by a single operator. Clinical success will be evaluated at 7 days, 1 month, and 3 months based on absence of pain, swelling, tenderness to percussion, and radiographic signs of periapical pathology.

ELIGIBILITY:
Inclusion Criteria:

* Mature permanent single rooted teeth with:

  * Symptomatic irreversible pulpitis
  * Age group 20-50 years

Exclusion Criteria:

* • Uncontrolled pulp heamorrhage (more than 5mins)

  * Necrotic pulp
  * Periapical periodontitis
  * Sinus tract
  * Abnormal tooth mobility
  * Single rooted teeth with internal or external root resorption
  * Calcified root canals

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Success of Complete Pulpotom | Evaluated at 7 days, 1 month, and 3 months post-procedure
  Clinical assessment of pain, swelling, and tenderness on percussion.
  Radiographic evaluation for absence of periapical lesions and root resorption.
  Success defined as absence of symptoms and radiographic signs of pathology, indicating maintenance of pulp vitality.

CONTACTS AND LOCATIONS:
Locations (1):
- Dental hospial, Hitec-IMS, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramani A, Sangwan P, Tewari S, Duhan J, Mittal S, Kumar V. Comparative evaluation of complete and partial pulpotomy in mature permanent teeth with symptomatic irreversible pulpitis: A randomized clinical trial. Int Endod J. 2022 May;55(5):430-440. doi: 10.1111/iej.13714. Epub 2022 Mar 10. PMID 35226769